CLINICAL TRIAL: NCT06922838
Title: Effectiveness of a Virtual Reality-based Multisensory Intervention for Postoperative Recovery in Patients Receiving Gynecological Surgery
Brief Title: The Effectiveness of a Virtual Reality-based Multisensory Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weifang Medical University (Other)
Responsible Party: Principal Investigator, Jiang Liu, Research investigator, Weifang Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2025YX406
Record Dates: First submitted 2025-04-03; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Gynecological Disease
Keywords: Pain management; Virtual reality; Gynecology; Postoperative recovery
MeSH Terms: conditions — Genital Diseases, Female; Agnosia | interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VR-Aromatherapy group (Other): The VR-Aromatherapy group received virtual reality intervention combined with aromatherapy for 20 minutes postoperatively. The intervention was started by an investigator from the return of the patient to the ward.
  Interventions: Other: Virtual Reality intervention; Other: Aromatherapy
- Aromatherapy group (Other): The Aromatherapy group received lavender aromatherapy for 20 minutes postoperatively. The intervention was started by an investigator from the return of the patient to the ward.
  Interventions: Other: Aromatherapy
- VR group (Other): The VR group received virtual reality intervention for 20 minutes postoperatively. The intervention was started by an investigator from the return of the patient to the ward.
  Interventions: Other: Virtual Reality intervention

INTERVENTIONS:
Other: Virtual Reality intervention — The head-mounted virtual reality device is used to provide patients with relaxing videos of nature scenes accompanied by calming music and guided meditations.
  Other Names: VR intervention
  Arms: VR group; VR-Aromatherapy group
Other: Aromatherapy — The cotton ball soaked in lavender essential oil is placed near the patient's pillow.
  Arms: Aromatherapy group; VR-Aromatherapy group

SUMMARY:
This study explores the effectiveness of a virtual reality-based multisensory intervention for postoperative recovery in patients receiving gynecological surgery.

DETAILED DESCRIPTION:
This study explores the effectiveness of a virtual reality-based multisensory intervention for postoperative recovery in patients receiving gynecological surgery. The results of the study included postoperative pain response, comfort, and anxiety of the patients.

ELIGIBILITY:
Inclusion Criteria: 1) significant postoperative pain response (VAS score over 4); 2) age greater than 18 years and volunteered to participate in this study.

Exclusion Criteria: 1) patients with psychosomatic disorders such as delirium, schizophrenia, and bipolar disorder; 2) patients with epilepsy, motion sickness, lightsensitivity, or other neurological diseases may have difficulty wearing the VR headset; 3) patients have severe heart, liver, kidney, blood, digestive, and nervous diseases.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study population was the patients undergoing gynecologic surgery.
Enrollment: 100 (Estimated)
Dates: Start 2025-04-06 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Pain response | The pain response of patients was assessed at 0.5 hour, 3 hour, 6 hour, 12 hour, 24 hour postoperatively, and immediately after intervention.
  The Visual Analog Scale (VAS) scale was used to assess the pain response of patients.
Anxiety | The anxiety level of patients was assessed immediately after the intervention.
  The Beck Anxiety Inventory (BAI) scale was used to assess the anxiety of patients.
Sleep quality | The sleep quality of patients was assessed at 24 hour postoperatively.
  The Pittsburgh Sleep Quality Index (PSQI) scale was used to assess the postoperative sleep quality of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Liu, M.D, Principal Investigator — Weifang Medical University